CLINICAL TRIAL: NCT02801097
Title: A Phase I, Open-Label, Multiple Ascending Dose Study to Assess the Safety and Tolerability of RRx-001 in Combination With Irinotecan in Metastatic or Advanced Cancer Patients Without Life-Prolonging Therapies of Demonstrated Clinical Benefit (PAYLOAD)
Brief Title: RRx-001 in Combination With Irinotecan in Metastatic or Advanced Cancer (PAYLOAD)
Acronym: PAYLOAD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sufficient patients enrolled to end study
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRx001-16-01
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Malignant Solid Tumor; Metastatic Cancer; Advanced Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — RRx-001; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RRx-001 + Irinotecan (Experimental): Cohorts of participants with an advanced, malignant, solid tumor(s) will receive weekly doses of RRx-001 for 3 weeks, switching at week 4 to every-other-week treatments of RRx-001 with irinotecan.
  Interventions: Drug: RRx-001; Drug: Irinotecan

INTERVENTIONS:
Drug: RRx-001
Drug: Irinotecan

SUMMARY:
This is a phase 1 open-label trial to evaluate the safety, pharmacodynamics and clinical activity of RRx-001 administered in combination with irinotecan.

RRx-001 is associated with resensitization to irinotecan in tumors that are previously refractory. This effect has been attributed to the ability of RRx-001 to restore the expression of aberrantly silenced genes, thus re-establishing pathway functions. However, resensitization may have more than one mechanism, among them Pgp pump inhibition and vascular modulation, leading to improved penetration of standard chemotherapy.

DETAILED DESCRIPTION:
This dose escalation study consists of 5 sequential dose cohorts each administered RRx-001 with irinotecan. After the first 3 subjects of each cohort complete Cycle 1, the safety will be assessed before moving to the next dose level. Subjects in the current cohort will continue treatment immediately following the completion of Cycle 1, for as long as therapy is tolerated and the RECIST v.1.1 definition of progression is not met.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of an advanced, malignant, solid tumor(s) with all standard treatment options having been exhausted or declined.
* Eastern Cooperative Group (ECOG) performance status is 0-2 at Screening.
* Measurable disease per RECIST v1.1 by radiographic techniques
* Acceptable liver function, serum creatinine and hematological status
* Female subjects of childbearing potential, and male subjects with partners of childbearing potential, must agree to use medically acceptable methods of contraception beginning on Study Day 1 and continuing until at least four weeks after administration of the subject's final dose of RRx-001.
* Subjects with brain metastases are eligible

Exclusion Criteria:

* Concurrent anticancer therapy; however, radiotherapy is allowed
* Any history of hypersensitivity to irinotecan
* Cholangitis that required treatment or intervention within 4 weeks of study enrollment
* Bilirubin > 2.0 mg/dL
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* If female, subject is pregnant and/or breastfeeding.
* UGT1A1*28 homozygote or heterozygote
* BMI >35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Number, frequency and type of adverse events | 14 Weeks

SECONDARY OUTCOMES:
Duration of clinical benefit rate | 1 year
  Duration of clinical benefit (Stable disease or better) using Response Evaluation Criteria in Solid Tumors [RECIST v1.1] criteria
Progression-Free Survival | 1 year
  Progression-Free Survival (PFS) using Response Evaluation Criteria in Solid Tumors
Overall Response rate | 1 year
  Proportion of patients with reduction in tumor burden using Response Evaluation Criteria in Solid Tumors
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Oronsky, MD, Study Director — EpicentRx, Inc.
Locations (2):
- United States (2):
  - University of California, Davis, Sacramento, California
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No